CLINICAL TRIAL: NCT03804320
Title: Sorveglianza Attiva Dei Tumori Renali T1a Uguali o Inferiori a 2 cm
Brief Title: Protocol Active Surveillance Small Renal Masses (SRMs)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Roberto Bertini, Principal investigator, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocollo SRM Sorv Attiva
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Kidney Cancer
Keywords: Kidney cancer; Active surveillance; Small renal masses; Partial nephrectomy
MeSH Terms: conditions — Kidney Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with small renal masses (Other): Active surveillance
  Interventions: Other: Active Surveillance

INTERVENTIONS:
Other: Active Surveillance

SUMMARY:
Prospective study of active surveillance, non-randomized, multicentric, in asymptomatic patients over the age of 50 years, not affected by other tumors, with occasional diagnosis of single monolateral solid renal mass equal to or less than 2 cm of diameter. Diagnosis will be performed with chest CT abdomen with contrast and / or MRI abdomen with Gadolinium (Gd); during the first year of active surveillance, the patient's status will be evaluated at 3, 6, 9 and 12 months from the diagnosis and, subsequently, according to the schedule of events shown in the table "Event Planning" At the end of the 5 years of follow up, the patient will be entrusted to his / her own treating physician, with indication to perform abdomen and chest x-ray echography every 6 months and thoracic abdomen TAC with contrast and / or MRI abdomen with (Gd) every 2 years up to 10 years from instrumental radiological diagnosis and registration and communication of the possible date of death and cause The primary caregivers and the patient will be contacted annually by the promoter center of the study at the end of the first 5 years of study follow up and the data will be entered in the database by the promoter center. The indication to surgical treatment or ablative treatment will be considered in the following cases: 1. appearance of metastasis 2. increase of the maximum diameter of the renal mass equal to or greater than 4 cm 3. time of doubling of the tumor mass size less than or equal to 12 months 4. appearance of symptoms associated with renal disease (pain, haematuria) 5. appearance of paraneoplastic syndrome (fever, cachexia, hypercalcemia, polycythemia, ranulocytosis) 6. willingness expressed by the patient to undergo surgery or ablative operation In the presence of at least one of the aforementioned criteria, the attending physician can evaluate the possible execution of renal biopsy. The finding of renal biopsy proved negative for neoplasia may allow the continuation of the active surveillance procedure undertaken, independently indi - ding from the presence of one of the above mentioned criteria. If the renal biopsy is negative, the therapeutic decision (continuation of the follow up within the protocol in question, surgery or exit from the protocol) will be agreed between the patient and the patient. In the case of a positive renal biopsy for renal neoplasia, the patient may be a candidate for renal tumorectomy / radical nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. ability to read, understand and interpret an informed consent;
2. voluntary subscription of the active surveillance protocol through written informed consent; 3) age over 50 years;

4) diagnosis of monolateral, monofocal, and first-rate solid renal mass less than 2 cm; 5) absence of symptoms due to renal tumor pathology.

Exclusion Criteria:

1. patients with a history of previous renal neoplasia;
2. monorenal patients;
3. patients with hereditary renal tumors (such as tuberous sclerosis and Von Hippel Lindau syndrome, etc.);
4. patients with metastasis;
5. patients suffering from immunodepressive diseases;
6. patients on concomitant therapy with chemotherapeutic agents or systemic immunosuppressants;
7. patients with life expectancy of less than 1 year.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-04-29 (Actual); Primary Completion 2023-12-11 (Estimated); Study Completion 2028-12-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate the therapeutic efficacy of active surveillance for small renal masses | 10 years
  Evaluate the therapeutic efficacy of active surveillance in patients with diagnosis of small renal tumor masses equal to or less than 2 cm in diameter.
Evaluate the proportion of patients who do not undergone active treatment | 10 years
  Proportion of patients who do not perform tumorectomy , tumor ablation or nephrectomy on the number of eligible patients that have been monitored for 12 months or more or have undergone surgery within 12 months

SECONDARY OUTCOMES:
Incidence and nature of disease progression during the period active surveillance | 10 years
  Determine the incidence and nature of disease progression during the period of active surveillance; determine the annual growth rate of SRMs equal to or less than 2 cm of diameter; evaluate the appearance of symptoms associated with the disease (pain, haematuria) or syndrome paraneoplasty (fever, cachexia, hypercalcemia, polycythemia, granulocytosis); establish possible factors clinical, pathological and biological predictive of local or metastatic disease progression or that require surgery.
Evaluation of disease progression | 10 years
  The disease progression is defined as the growth of the maximum diameter of the renal mass equal to or more than 4 cm or doubling the tumor volume over a period of time ≤ 12 months. It is considered sign of progression also the vascular invasion, with the appearance of thrombosis of the renal vein or of the inferior vena cava;

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Bertini, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Volpe A, Panzarella T, Rendon RA, Haider MA, Kondylis FI, Jewett MA. The natural history of incidentally detected small renal masses. Cancer. 2004 Feb 15;100(4):738-45. doi: 10.1002/cncr.20025. PMID 14770429
- [Background] Lane BR, Abouassaly R, Gao T, Weight CJ, Hernandez AV, Larson BT, Kaouk JH, Gill IS, Campbell SC. Active treatment of localized renal tumors may not impact overall survival in patients aged 75 years or older. Cancer. 2010 Jul 1;116(13):3119-26. doi: 10.1002/cncr.25184. PMID 20564627
- [Background] Tada S, Yamagishi J, Kobayashi H, Hata Y, Kobari T. The incidence of simple renal cyst by computed tomography. Clin Radiol. 1983 Jul;34(4):437-9. doi: 10.1016/s0009-9260(83)80238-4. PMID 6872451
- [Background] Lane BR, Chen H, Morrow M, Anema JG, Kahnoski RJ. Increasing use of kidney sparing approaches for localized renal tumors in a community based health system: impact on renal functional outcomes. J Urol. 2011 Oct;186(4):1229-35. doi: 10.1016/j.juro.2011.05.081. Epub 2011 Aug 17. PMID 21849192
- [Background] Thompson RH, Kaag M, Vickers A, Kundu S, Bernstein M, Lowrance W, Galvin D, Dalbagni G, Touijer K, Russo P. Contemporary use of partial nephrectomy at a tertiary care center in the United States. J Urol. 2009 Mar;181(3):993-7. doi: 10.1016/j.juro.2008.11.017. Epub 2009 Jan 16. PMID 19150552
- [Background] Dulabon LM, Lowrance WT, Russo P, Huang WC. Trends in renal tumor surgery delivery within the United States. Cancer. 2010 May 15;116(10):2316-21. doi: 10.1002/cncr.24965. PMID 20225227
- [Background] Campbell SC, Novick AC, Belldegrun A, Blute ML, Chow GK, Derweesh IH, Faraday MM, Kaouk JH, Leveillee RJ, Matin SF, Russo P, Uzzo RG; Practice Guidelines Committee of the American Urological Association. Guideline for management of the clinical T1 renal mass. J Urol. 2009 Oct;182(4):1271-9. doi: 10.1016/j.juro.2009.07.004. Epub 2009 Aug 14. No abstract available. PMID 19683266
- [Background] Klinghoffer Z, Tarride JE, Novara G, Ficarra V, Kapoor A, Shayegan B, Braga LH. Cost-utility analysis of radical nephrectomy versus partial nephrectomy in the management of small renal masses: Adjusting for the burden of ensuing chronic kidney disease. Can Urol Assoc J. 2013 Mar-Apr;7(3-4):108-13. doi: 10.5489/cuaj.502. PMID 23671525
- [Background] Lane BR, Babineau D, Kattan MW, Novick AC, Gill IS, Zhou M, Weight CJ, Campbell SC. A preoperative prognostic nomogram for solid enhancing renal tumors 7 cm or less amenable to partial nephrectomy. J Urol. 2007 Aug;178(2):429-34. doi: 10.1016/j.juro.2007.03.106. Epub 2007 Jun 11. PMID 17561141
- [Background] Remzi M, Ozsoy M, Klingler HC, Susani M, Waldert M, Seitz C, Schmidbauer J, Marberger M. Are small renal tumors harmless? Analysis of histopathological features according to tumors 4 cm or less in diameter. J Urol. 2006 Sep;176(3):896-9. doi: 10.1016/j.juro.2006.04.047. PMID 16890647
- [Background] Frank I, Blute ML, Cheville JC, Lohse CM, Weaver AL, Zincke H. Solid renal tumors: an analysis of pathological features related to tumor size. J Urol. 2003 Dec;170(6 Pt 1):2217-20. doi: 10.1097/01.ju.0000095475.12515.5e. PMID 14634382
- [Background] Volpe A, Cadeddu JA, Cestari A, Gill IS, Jewett MA, Joniau S, Kirkali Z, Marberger M, Patard JJ, Staehler M, Uzzo RG. Contemporary management of small renal masses. Eur Urol. 2011 Sep;60(3):501-15. doi: 10.1016/j.eururo.2011.05.044. Epub 2011 Jun 1. PMID 21664040
- [Background] Hollingsworth JM, Miller DC, Daignault S, Hollenbeck BK. Rising incidence of small renal masses: a need to reassess treatment effect. J Natl Cancer Inst. 2006 Sep 20;98(18):1331-4. doi: 10.1093/jnci/djj362. PMID 16985252
- [Background] Raj GV, Thompson RH, Leibovich BC, Blute ML, Russo P, Kattan MW. Preoperative nomogram predicting 12-year probability of metastatic renal cancer. J Urol. 2008 Jun;179(6):2146-51; discussion 2151. doi: 10.1016/j.juro.2008.01.101. Epub 2008 Apr 18. PMID 18423735
- [Background] Smaldone MC, Kutikov A, Egleston BL, Canter DJ, Viterbo R, Chen DY, Jewett MA, Greenberg RE, Uzzo RG. Small renal masses progressing to metastases under active surveillance: a systematic review and pooled analysis. Cancer. 2012 Feb 15;118(4):997-1006. doi: 10.1002/cncr.26369. Epub 2011 Jul 15. PMID 21766302
- [Background] Nguyen MM, Gill IS. Effect of renal cancer size on the prevalence of metastasis at diagnosis and mortality. J Urol. 2009 Mar;181(3):1020-7; discussion 1027. doi: 10.1016/j.juro.2008.11.023. Epub 2009 Jan 16. PMID 19150563
- [Background] Jewett MA, Mattar K, Basiuk J, Morash CG, Pautler SE, Siemens DR, Tanguay S, Rendon RA, Gleave ME, Drachenberg DE, Chow R, Chung H, Chin JL, Fleshner NE, Evans AJ, Gallie BL, Haider MA, Kachura JR, Kurban G, Fernandes K, Finelli A. Active surveillance of small renal masses: progression patterns of early stage kidney cancer. Eur Urol. 2011 Jul;60(1):39-44. doi: 10.1016/j.eururo.2011.03.030. Epub 2011 Apr 1. PMID 21477920
- [Background] Mason RJ, Abdolell M, Trottier G, Pringle C, Lawen JG, Bell DG, Jewett MA, Klotz L, Rendon RA. Growth kinetics of renal masses: analysis of a prospective cohort of patients undergoing active surveillance. Eur Urol. 2011 May;59(5):863-7. doi: 10.1016/j.eururo.2011.02.023. Epub 2011 Feb 22. PMID 21353376
- [Background] Ozsoy M, Klatte T, Waldert M, Remzi M. Surveillance for the management of small renal masses. Adv Urol. 2008;2008:196701. doi: 10.1155/2008/196701. PMID 18704192
- [Background] Patel N, Cranston D, Akhtar MZ, George C, Jones A, Leiblich A, Protheroe A, Sullivan M. Active surveillance of small renal masses offers short-term oncological efficacy equivalent to radical and partial nephrectomy. BJU Int. 2012 Nov;110(9):1270-5. doi: 10.1111/j.1464-410X.2012.11130.x. Epub 2012 May 4. PMID 22564495
- [Background] Barrisford GW, Singer EA, Rosner IL, Linehan WM, Bratslavsky G. Familial renal cancer: molecular genetics and surgical management. Int J Surg Oncol. 2011;2011:658767. doi: 10.1155/2011/658767. Epub 2011 Aug 22. PMID 22312516
- [Background] Walther MM, Choyke PL, Glenn G, Lyne JC, Rayford W, Venzon D, Linehan WM. Renal cancer in families with hereditary renal cancer: prospective analysis of a tumor size threshold for renal parenchymal sparing surgery. J Urol. 1999 May;161(5):1475-9. doi: 10.1016/s0022-5347(05)68930-6. PMID 10210376
- [Background] Ayati M, Nikfallah A, Jabalameli P, Najjaran Tousi V, Noroozi M, Jamshidian H. Extensive surgical management for renal tumors with inferior vena cava thrombus. Urol J. 2006 Fall;3(4):212-5. PMID 17559043
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716